CLINICAL TRIAL: NCT04569916
Title: An Exploratory Study to Evaluate Radiotherapy Combined With Irinotecan Liposome and Apatinib Followed by PD-1 Antibody and Apatinib for the Treatment of Advanced Solid Tumors That Failed Standard Treatments
Brief Title: Radiotherapy Combined With Irinotecan and Apatinib Followed by PD-1 Antibody and Apatinib for Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Baorui Liu, chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-RT-IRI-SHR1210-APA
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Radiotherapy; irinotecan sucrosofate; apatinib; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): radiotherapy combined with irinotecan liposome and apatinib followed by PD-1 antibody and apatinib
  Interventions: Radiation: radiotherapy; Drug: irinotecan liposome; Drug: apatinib; Drug: PD-1 antibody

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy combined with irinotecan liposome and apatinib followed by PD-1 antibody and apatinib
Drug: irinotecan liposome — radiotherapy combined with irinotecan liposome and apatinib followed by PD-1 antibody and apatinib
Drug: apatinib — radiotherapy combined with irinotecan liposome and apatinib followed by PD-1 antibody and apatinib
  Other Names: Apatinib Mesylate Tablets
Drug: PD-1 antibody — radiotherapy combined with irinotecan liposome and apatinib followed by PD-1 antibody and apatinib

SUMMARY:
An exploratory study to evaluate for the treatment of advanced solid tumors that failed standard treatments.

DETAILED DESCRIPTION:
This is a prospective, single-arm, observational study. After the subjects meet the inclusive and exclusive criteria, then they will receive radiotherapy combined with irinotecan liposome and apatinib followed by PD-1 antibody and apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old, both men and women;
2. Eastern Cooperative Oncology Group performance status 0-1;
3. Pathologically confirmed recurrent or metastatic solid tumors (pancreatic cancer, colorectal cancer, non-small cell lung cancer, hepatocellular carcinoma, head and neck tumors, gastric cancer, etc.) that failed, couldn't tolerate or lacked standard treatments;
4. According to the response evaluation criteria in solid tumor (RECIST 1.1), at least two measurable lesion for radiotherapy; for patients with brain metastases, there must be at least one metastasis outside the brain;
5. Expected survival period ≥ 12 weeks;
6. The main organ function and bone marrow function are normal, meeting the following requirements:

   1. Hemoglobin ≥ 90 g / L; (No blood transfusion within 14 days)
   2. Absolute neutrophil count ≥1.5×109/L;
   3. platelet count ≥ 90 × 109 / L;
   4. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
   5. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN; if there is liver metastasis, ALT and AST ≤ 5 times ULN;
   6. creatinine ≤ 1.5 times ULN;
   7. Left ventricular ejection fraction (LVEF) ≥ 50%; QTc male <450ms, female <470ms;
7. Patients who have not received anticoagulant therapy have an international normalized ratio (INR) of ≤1.5 and partial thromboplastin time (APTT) ≤1.5 times ULN. Patients receiving total or parenteral anticoagulant therapy should be stable for at least 2 weeks before entering the clinical study, and the results of the coagulation test are within the limits of local treatment;
8. Women of childbearing age must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment, and voluntarily use the appropriate method for contraception during the observation period and within 3 months after the last administration of the study drug; for men, surgical sterilization or consent to use appropriate methods of contraception during the observation period and within 3 months after the last administration of the study drug.
9. The toxicity of receiving pre-treatment has been restored to ≤grade 1 (if the patient received surgery, the wound should be completely healed);
10. Patients voluntarily participate in and sign informed consent, and they are expected to have good compliance and can cooperate with the research according to the program requirements.

Exclusion Criteria:

1. Received any kind of anti-tumor treatment within 4 weeks before enrollment, including radiotherapy, chemotherapy, molecular targeted therapy, and immunotherapy, or participate in another interventional clinical trial;
2. Major surgery was performed within 4 weeks before enrollment (except for minor surgery, such as placement of vascular access); surgical fixation of the bone lesions to be irradiated is required, and mechanical stabilization is indicated;
3. There is a third interstitial fluid (such as a large amount of pleural effusion or ascites) that has clinical symptoms and cannot be controlled by drainage or other methods;
4. Even after medical treatment, hypertension is still poorly controlled (continuous increase in systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg)
5. Suffering from uncontrolled clinical symptoms or diseases of the heart, such as (1) New York Heart Association II and above heart failure; (2) unstable angina; (3) myocardial infarction within 1 year; (4) clinically significant patients with supraventricular or ventricular arrhythmia requiring clinical intervention;
6. Patients with any active autoimmune disease or history of autoimmune disease, including interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, and hypothyroidism (hypothyroidism can be included after hormone replacement therapy), except for patients with vitiligo or childhood asthma that has been completely relieved and does not require any intervention after adulthood. Asthma that requires intermittent use of bronchodilators or other medical intervention should also be excluded.
7. People with congenital or acquired immune function defects, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA is higher than the lower limit of the analytical method) or co-infection with hepatitis B and C;
8. Severe infection within 4 weeks before the first dose (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever >38.5 °C during screening/before first dose;
9. Events of arterial or venous thrombosis occurring within 6 months before enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
10. Have had or have other systemic malignancies in the last 5 years (except for cured skin basal cell carcinoma and cervical carcinoma in situ and ovarian cancer);
11. Those who are known to be allergic to any study drug;
12. Pregnant patients, lactating patients, or patients with reproductive ability are not willing to take effective contraceptive measures;
13. Have a clear history of neurological or mental disorders, including epilepsy and dementia;
14. Known uncontrolled or symptomatic active central nervous system (CNS) metastases, manifested by clinical signs, cerebral edema, spinal cord compression, cancerous meningitis, pia mater disease, and/or progressive growth;
15. Patients who are unable to swallow the study drug, such as patients with chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis), intestinal obstruction, and other various factors that affect drug administration and absorption;
16. Other circumstances that the investigator believes are not suitable for inclusion. If accompanied by family or social factors, it will affect the safety of the subject or the collection of data and samples.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard

SECONDARY OUTCOMES:
Disease Control Rate | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Clinical benefit rate | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Correlation between immune microenvironment parameters of target lesions and efficacy | 2 years
  Evaluated by researchers based on the RECIST 1.1 standard
Drug-related Adverse Event | 2 years
  Evaluated by researchers
Drug-related Serious Adverse Event | 2 years
  Evaluated by researchers

CONTACTS AND LOCATIONS:
Overall Officials: Baorui Baorui Liu, Doctor, Principal Investigator — Nanjing Drum Tower Hospital, The Affiliated of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, The Affiliated of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Shen J, Yan J, Du J, Li X, Wei J, Liu Q, Yong H, Wang X, Chang X, Ding Z, Sun W, Liu C, Zhu S, Guo J, Li H, Liu Y, Zhang W, Liu Z, Li R, Liu B. Multicenter, single-arm, phase II study (CAP) of radiotherapy plus liposomal irinotecan followed by camrelizumab and anti-angiogenic treatment in advanced solid tumors. Front Immunol. 2023 Mar 28;14:1133689. doi: 10.3389/fimmu.2023.1133689. eCollection 2023. PMID 37056765